CLINICAL TRIAL: NCT03347214
Title: dbGaP Protocol: The Pediatric Cardiac Genetics Consortium (PCGC)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918006; 18-H-N006
Record Dates: First submitted 2017-11-17; First posted 2017-11-20 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Congenital Heart Disease
Keywords: dbGaP
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: People who already participated in the Pediatric Cardiac Genomics Consortium (PCGC) study

SUMMARY:
Background:

Researchers do not know much about the causes of congenital heart disease (CHD). They do know that many factors play a role. Some factors are environmental. Some are genetic. But few specific factors have been identified. And researchers do not know how many involve genes. They want to study data that has already been collected from people with CHD and their families.

Objectives:

To identify genetic variations related to CHD. To study molecules related to vascular disease in order to learn new ways to treat it.

Eligibility:

People who already participated in the Pediatric Cardiac Genomics Consortium (PCGC) study

Design:

Researchers will study data that was already collected in the PCGC. There will be no active participants.

Researchers will get access to the data through the coordinating center. They will not download data to local storage devices.

The data will have no personally identifying information....

DETAILED DESCRIPTION:
Current understanding of the causes of congenital heart disease (CHD) is limited, but CHD is known to be multifactorial and affected by a combination of environmental, teratogenic, and genetic causes. Furthermore, both genetic and environmental factors have been proposed to act as disease modifiers, accounting for a wide variation in phenotypic expression and clinical outcomes of these disorders. To date however, few specific genetic or environmental causative factors have been identified, nor is it even known what proportion of cases involve genetic factors.

ELIGIBILITY:
* Retrospective Analysis Study. Data will be analyzed from subjects from cardiovascular disease databases.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People who already participated in the Pediatric Cardiac Genomics Study
Sampling Method: Non-Probability Sample
Enrollment: 6260 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Identification of novel genetic variants associated with a CHD phenotype | Ongoing
  de novo variants, SNPs, and CNVs

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Kaltman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States